CLINICAL TRIAL: NCT07325773
Title: Effects of Magnesium Sulfate on Intraoperative Oxygenation and Lung Mechanics During One-Lung Ventilation: A Prospective Observational Study
Brief Title: Effects of Magnesium Sulfate on Oxygenation and Lung Mechanics During One-Lung Ventilation
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, Associate Professor, Marmara University
Other Study IDs: 09.2025.463
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Intraoperative Oxygenation and Pulmonary Mechanics
Keywords: Magnesium Sulfate; One-Lung Ventilation; Lung Mechanics; Oxygenation; Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Magnesium Sulfate Group Label: Magnesium Sulfate Group: Patients receiving intravenous magnesium sulfate during the surgery as part of standard anesthetic management.
- Group 2 - Control Group Label: Control Group: Patients undergoing one-lung ventilation without the administration of magnesium sulfate

SUMMARY:
This prospective observational study aims to evaluate the effects of intravenous magnesium sulfate on intraoperative oxygenation and lung mechanics in patients undergoing thoracic surgery with one-lung ventilation. Magnesium sulfate has been reported to have potential bronchodilatory and anti-inflammatory properties, which may improve gas exchange and respiratory mechanics during lung isolation.

In this study, patients who receive magnesium sulfate as part of standard anesthetic management will be compared with those who do not receive the drug. Oxygenation parameters, dynamic and static lung mechanics, airway pressures, and ventilation-related indices will be recorded throughout the intraoperative period. The findings of this study may help clarify whether magnesium sulfate provides measurable respiratory benefits during one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 80 years Scheduled for elective thoracic surgery performed with video-assisted thoracoscopic surgery (VATS) requiring one-lung ventilation under general anesthesia.

ASA physical status II-III Ability to provide informed consent Undergoing general anesthesia with double-lumen tube placement

Exclusion Criteria:

* Patients undergoing pneumonectomy
* Patients with renal, hepatic, or cardiovascular failure
* Patients with a BMI < 15 kg/m² or > 35 kg/m²
* Patients with a preoperative pulmonary function test showing FEV₁ < 1.5 liters
* Patients who are transferred to the intensive care unit intubated in the postoperative period
* Patients with physical or mental conditions that prevent the performance of pulmonary function testing factors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients undergoing elective thoracic surgery performed with video-assisted thoracoscopic surgery (VATS) requiring one-lung ventilation under general anesthesia. The study population consists of individuals scheduled for minimally invasive lung resections or other VATS procedures necessitating lung isolation. Patients receiving magnesium sulfate intraoperatively and those not receiving it will be prospectively observed. Patients undergoing pneumonectomy, those with significant organ failure, extreme BMI values, or inadequate pulmonary function will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Change in Intraoperative Oxygenation (PaO₂/FiO₂ Ratio) | From induction of anesthesia to the end of one-lung ventilation (approximately 2-3 hours)
  The PaO₂/FiO₂ ratio will be measured to evaluate intraoperative oxygenation during the surgery. Measurements will be recorded after induction of anesthesia (baseline) and at predefined intraoperative time points. The primary outcome is the change in PaO₂/FiO₂ ratio between baseline and intraoperative measurements in patients receiving magnesium sulfate versus control.

SECONDARY OUTCOMES:
Changes in Airway Pressures (Peak and Plateau Pressures) | From induction of anesthesia to the end of one-lung ventilation (approximately 2-3 hours).
  Peak inspiratory pressure (PIP) and plateau pressure (Pplat) will be measured to assess changes in airway pressures during one-lung ventilation in patients receiving magnesium sulfate compared with control.
Dynamic Lung Compliance and Airway Resistance (Raw) | Intraoperative period (approximately 2-3 hours).
  Dynamic compliance (Cdyn) will be recorded at predefined intraoperative time points to evaluate changes in pulmonary mechanics associated with magnesium sulfate administration.Airway resistance (Raw) will be measured at predefined intraoperative time points using ventilator-derived data. Raw will be compared between patients receiving magnesium sulfate and those in the control group to assess the effect of magnesium sulfate on airway resistance during one-lung ventilation.
Postoperative Arterial Oxygen Partial Pressure (PaO₂) on Room Air | Within the first postoperative hour while breathing room air.
  Arterial oxygen partial pressure (PaO₂) will be measured in the postoperative period while patients are breathing room air. This outcome will be used to assess whether intraoperative magnesium sulfate administration has an effect on early postoperative oxygenation following one-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Meliha ORHON ERGÜN, Study Chair — Marmara University Faculty of Medicine, Department of Anesthesiology and Reanimation; İlayda AKARSU KAYA, Principal Investigator — Marmara University Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University Faculty of Medicine, Basibuyuk Campus, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No